CLINICAL TRIAL: NCT06719882
Title: A Prospective Study of Vivity & Vivity Toric IOL in Taiwan: Results and Analysis
Brief Title: Vivity Study in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: Taipei Nobel Eye Clinic (Other)
Responsible Party: Principal Investigator, Chao-Kai Chang, Doctor, Taipei Nobel Eye Clinic
Other Study IDs: 005
Record Dates: First submitted 2024-11-10; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cataract
Keywords: Intraocular lens; Extended depth of focus
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vivity/Vivity toric

SUMMARY:
The aim of study is to evaluate the quality of vision after bilateral Vivity or Vivity toric EDOF IOLs implantation in Taiwan.

DETAILED DESCRIPTION:
This study was a prospective, single arm study. The inclusion criteria for this study were the presence of cataracts in both eyes and corrected distance visual acuity (CDVA) of both eyes under 20/40, who received bilateral Vivity IOL implantation after cataract surgery, targeting emmetropia or mini-monovision of both eyes. Phacoemulsification cataract surgery was performed on all patients. The exclusion criteria were complicated cataract; corneal opacities or irregularities; severe dry eye (Schirmer's test I ≤ 5 mm); amblyopia; anisometropia; surgical complications such as posterior capsular bag rupture, vitreous loss, or IOL tilt/decentration; coexisting ocular pathologies such as glaucoma, nondilating pupil, history of intraocular surgery, refractive surgery, or retinopathy; optic nerve or macular diseases; and refusal or inability to maintain follow-up. When corneal astigmatism was more than 0.75 diopters (D), a toric IOL was implanted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age-related cataract requiring surgery treatment
* Patient who received bilateral, uneventful implantation of Vivity IOLs
* Patient's IOL power is between 10-30D, and T2-T6 for toric correction
* Cataract grade 0~3 based on the Wisconsin cataract grading system

  • Exclusion criteria:
* Cataract grade 4~5 based on the Wisconsin cataract grading system
* Patient's IOL power is outside of 10-30D or T2-T6 for toric correction
* Patient with the following ocular comorbidities:
* Corneal opacities or irregularities;
* Severe dry eye;
* Amblyopia;
* Glaucoma;
* Non-dilating pupil;
* History of intraocular surgery, laser therapy, or retinopathy;
* Optic nerve or macular diseases;
* Uncontrolled diabetic mellitus or systemic immune disease;
* Refusal or unable to maintain follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who intended for sequential bilateral cataract surgery and implanted with Vivity/Vivity IOL would be asked to include in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (LogMAR) | From enrollment to the end of treatment at 3 months
  Uncorrected binocular far, intermediate and near visual acuity. Corrected binocular far, intermediate and near visual acuity.

OTHER OUTCOMES:
Intermediate reading speed (seconds) | From enrollment to the end of treatment at 3 months
  The intermediate reading speed was measured by IReST - International Reading Speed Texts Chinese Edition

CONTACTS AND LOCATIONS:
Overall Officials: ChaoKai Chang, Ph.D., Study Director — Taiwan Nobel Eye Clinic
Locations (1):
- Taiwan Nobel Eye Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kandavel R, Colvard M, Dredge J, Bayle M, Alam T, Snyder J, Hall B. Comparative Study Between Non-Diffractive Extended Depth of Focus and Monofocal Intraocular Lenses. Clin Ophthalmol. 2023 Apr 14;17:1161-1168. doi: 10.2147/OPTH.S402069. eCollection 2023. PMID 37082300
- [Result] Hovanesian JA, Jones M, Allen Q. The Vivity Extended Range of Vision IOL vs the PanOptix Trifocal, ReStor 2.5 Active Focus and ReStor 3.0 Multifocal Lenses: A Comparison of Patient Satisfaction, Visual Disturbances, and Spectacle Independence. Clin Ophthalmol. 2022 Jan 18;16:145-152. doi: 10.2147/OPTH.S347382. eCollection 2022. PMID 35082481